CLINICAL TRIAL: NCT04909333
Title: Exenatide-test for Diagnosing Endogenous Hyperinsulinemic Hypoglycemia
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Gottfried und Julia Bangerter- Rhyner-Stiftung, Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020-00169; qu20Antwi2
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Endogenous Hyperinsulinism
Keywords: fasting test; Blood glucose; insulin; proinsulin; C-peptide; betahydroxybutyrate; hypoglycemia
MeSH Terms: conditions — Hyperinsulinism; Insulin Resistance; Diabetes Mellitus, Insulin-Dependent, 2; Hypoglycemia | interventions — Exenatide; Saline Solution

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, cross-over, placebo controlled pilot, proof of principle clinical study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (EHH Patients) (Experimental): Group A will receive a placebo injection (0.9% saline solution) on Day 1 and 10μg Exenatide injection on Day 2.
  Interventions: Drug: Exenatide; Drug: 0.9% saline solution
- Group B (EHH Patients) (Experimental): Group B will receive a 10μg Exenatide injection on Day 1 and placebo injection (0.9% saline solution) on Day 2.
  Interventions: Drug: Exenatide; Drug: 0.9% saline solution
- Group C (control subjects) (Experimental): Control subjects without evidence for EHH defined by no glucose levels below 3.0 mmol/l during a 7-day CGFS (Freestyle libre) and matched to EHH patients for age, gender and BMI will receive only on one study day a single intravenous injection of 10μg Exenatide and compared to group A patients on Day 2. They will not receive a Placebo injection.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Day1: After a standardized night meal (Maizena 40g plus dessert) at 22 p.m. on the day before, patients receive Exenatide study medication according to the randomization list (injection done slowly over 2 min.). Regular clinical examination of vegetative and neurological state will be done as well as continuous blood sugar measurements and blood withdrawals will be performed.
  Day2:
  The procedure is equal to study day 1. Instead of Exenatide, a 10ml 0.9% saline solution will be administered intravenously.
  Other Names: Day 1 Exenatide; Day 2 : 0.9% saline solution
Drug: 0.9% saline solution — Day1: After a standardized night meal (Maizena 40g plus dessert) at 22 p.m. on the day before, patients receive 0.9% saline solution according to the randomization list (injection done slowly over 2 min.). Regular clinical examination of vegetative and neurological state will be done as well as continuous blood sugar measurements and blood withdrawals will be performed.
  Day2:
  The procedure is equal to study day 1. Instead of 0.9% saline solution, Exenatide will be administered intravenously.
  Other Names: Day 1 : 0.9% saline solution, Day 2 Exenatide
  Arms: Group A (EHH Patients); Group B (EHH Patients)

SUMMARY:
This study is to evaluate the concept of the exenatide test for diagnosis of EHH (earlier induction of symptomatic hypoglycemia compared to placebo within 4 hours after injection).

DETAILED DESCRIPTION:
Endogenous hyperinsulinemic hypoglycemia (EHH) is defined as inappropriate endogenous insulin secretion leading to hypoglycemia and associated symptoms. The most frequent diagnosis is an insulin-secreting pancreatic neuroendocrine tumor, but other diagnoses such as nesidioblastosis of the pancreatic islets are also possible. Biochemically, EHH is characterized by low glucose concentrations in the presence of inappropriately increased C-peptide (endogenous insulin secretion) and insulin levels. The conventional fasting test is at present the gold standard to document EHH.

Radiolabeled Exenatide for localizing insulinomas in patients with biochemically proven EHH has been evaluated and an exenatide-test in an outpatient setting may be able to replace the fasting test, by an early symptomatic hypoglycemia compared to a prolonged inpatient monitoring.

This study is to investigate the concept of the exenatide test to diagnose EHH.

ELIGIBILITY:
Patients with suspicion for an insulinoma fulfilling all of the following inclusion criteria are eligible for the study:

Inclusion Criteria:

* Informed Consent as documented by signature
* Biochemically proven endogenous hyperinsulinemic hypoglycemia: neuroglycopenic symptoms in the fasting state with low plasma glucose, inappropriately high serum insulin and C-peptide concentrations (standardized 72h fasting test).).

Participants as control subjects fulfilling all of the following inclusion criteria are eligible for the study:

Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Possession of the adequate match criteria (age, BMI and gender) to patients with suspicion for an insulinoma

Exclusion Criteria:

* Known hypersensitivity or allergy to Exenatide
* Pregnant or breastfeeding female patients. A pregnancy test will be performed in all women of child bearing potential.
* Calculated creatinine clearance below 40 ml/min
* No signed informed consent
* Intake of any glucagon-like peptide (GLP)-1 analogue (such as Byetta® or Bydureon®[= Exenatide])
* prediabetes or diabetes (HbA1c > 5.7 %)
* Previous abdominal surgery in the gastrointestinal tract
* Any concomitant glucose-lowering drug (i. e. insulin, sulfonyl urea)
* Any known intolerance to standardized meal (Maizena)
* Any uncontrolled significant medical, psychiatric or surgical condition (active infection, unstable angina pectoris, cardiac arrhythmia, poorly controlled hypertension, uncontrolled congestive heart disease, etc.) or laboratory findings that might jeopardize the patient's safety or that would limit compliance with the objectives and assessments of the study.
* Any mental conditions which prevent the patient from understanding the type, extent and possible consequences of the study and/or an uncooperative attitude from the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
time to symptomatic hypoglycemia after exenatide test compared to placebo | within 4 hours after injection
  time to symptomatic hypoglycemia after exenatide test compared to placebo

SECONDARY OUTCOMES:
time dependent decrease (time Δ from injection in min) of blood glucose (% or mmol/l)) | within 4 hours after injection
  time dependent decrease (time Δ from injection in min) of blood glucose (% or mmol/l)) that can best discriminate from placebo injection
time to symptoms | within 4 hours after injection
  time to symptoms of the exenatide test in comparison to the placebo injection of 10ml 0.9% saline solution
time to hypoglycemia (time to reach blood sugar level ≤ 2.5 mmol/l) in the exenatide test in comparison to the placebo | within 4 hours after injection
  time to hypoglycemia (time to reach blood sugar level ≤ 2.5 mmol/l) in the exenatide test in comparison to the placebo
time to hypoglycemia (time to reach blood sugar level ≤ 2.5 mmol/l) in the exenatide test in comparison to the fasting test | within 4 hours after injection
  time to hypoglycemia (time to reach blood sugar level ≤ 2.5 mmol/l) in the exenatide test in comparison to the fasting test
time to symptoms in the exenatide test in comparison to the fasting test | within 4 hours after injection
  time to symptoms in the exenatide test in comparison to the fasting test
change in levels of plasma glucose compared to placebo compared to placebo | within 4 hours after injection
  change in levels of plasma glucose compared to placebo
change in levels of insulin compared to placebo | within 4 hours after injection
  change in levels of insulin compared to placebo
change in levels of C-peptide compared to placebo | within 4 hours after injection
  change in levels of C-peptide compared to placebo compared to placebo
change in levels of proinsulin compared to placebo | within 4 hours after injection
  change in levels of proinsulin compared to placebo
change in levels of ß-hydroxybutyrate compared to placebo | within 4 hours after injection
  change in levels of ß-hydroxybutyrate compared to placebo
costs of exenatide test setting (CHF) | within 4 hours after injection
  Comparison of costs of exenatide test setting with fasting test setting

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Christ, Prof. Dr. med., Study Director — University Hospital of Basel, Interdisciplinary Endocrinology
Locations (1):
- University Hospital Basel, Division of Nuclear Medicine, Basel, Switzerland

REFERENCES:
- [Derived] Hepprich M, Romberg C, Mudry J, Refardt J, Wild D, Antwi K, Christ E. Exenatide for diagnosing endogenous hyperinsulinemic hypoglycemia: a randomized placebo-controlled, double-blind, cross-over proof-of-principle study. Eur J Endocrinol. 2025 Jul 31;193(2):247-254. doi: 10.1093/ejendo/lvaf153. PMID 40747712